CLINICAL TRIAL: NCT06277700
Title: A Comparison of the Effectiveness of Dynamic Neuromuscular Stabilizatıon Exercises and Chiropractıc HVLALumbar Manipulatıon in Individuals with Chronic Non-specific Low Back Pain
Brief Title: Effects of Dynamic Stabilizatıon Exercises and HVLA Manipulatıon in Low Back Paın
Acronym: DNSHVLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SEFA HAKTAN HATIK (Other)
Responsible Party: Sponsor-Investigator, SEFA HAKTAN HATIK, Assistant Professor, Sinop University
Organization: Sinop University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CMT001
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-02

CONDITIONS: Low Back Pain; Neuromuscular Subluxation of Joint
Keywords: Spinal Manipulation; Dynamic Neuromuscular Stabilization; Low Back Pain; Posture; Non - spesific
MeSH Terms: conditions — Low Back Pain | interventions — Manipulation, Chiropractic

STUDY DESIGN:
Intervention Model Description: 60 people will participate in the study and the participants will be divided into four groups. The groups will be formed as chiropractic manipulation (CM) group (n=15), dynamic neuromuscular stabilization (DNS) group (n=15), CM + DNS group (n=15) and control group (CG) (n=15). Chiropractic manipulation will be performed once in the side-lying position. An individualized exercise program will be applied to the DNS group under the supervision of a physiotherapist. Kruskal Wallis test for comparisons of quantitative variables between 4 independent groups; Mann Whitney U test with Bonferonni correction will be used in double subgroup comparisons of significant variables. Friedman test was used for comparisons of quantitative variables in 3 dependent groups. Wilcoxon test with Bonferonni correction will be used for two-way subgroup comparisons for significant variables. In all statistical analyzes in the study, results with a p value below 0.05 will be considered statistically significant.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Chiropractic Manipulation (CM) Group (Experimental): In the side lying position, lumbar chiropractic manipulation will be performed over the transverse process of the vertebra thought to have vertebral subluxation. A total of 8 sessions of chiropractic manipulation will be performed 2 times a week.
  Interventions: Other: Chiropractic Manipulation (HVLA - high velocity low amplitude)
- Dynamic Neuromuscular Stabilization (DNS) Group (Experimental): Participants in the groups receiving DNS exercise therapy will be given individualized exercises under the supervision of a physiotherapist. Firstly, the participants will be taught the skill of posterior diaphragm activation in the supine position and the ability to direct the intra-abdominal pressure caudally, while preventing the cranial movement of the thorax, so that the chest and pelvis are in a neutral position and the thoracic diaphragm and pelvis are aligned in parallel. Our aim in this alignment is that with the correct diaphragm movement pattern, the deep stabilizers will be activated as a reflex response to intra-abdominal pressure change. Participants will be asked to focus on and maintain this alignment throughout the entire DNS exercise pattern. Exercises will be done 2 times a week for 50 minutes for 4 weeks.
  Interventions: Other: Dynamic Neuromuscular Stabilization
- CM + DNS Group (Experimental): This group receives a treatment as a combination of the treatments described above.
  Interventions: Other: Chiropractic Manipulation (HVLA - high velocity low amplitude); Other: Dynamic Neuromuscular Stabilization
- Control Group (No Intervention): No treatment will be applied to the control group.

INTERVENTIONS:
Other: Chiropractic Manipulation (HVLA - high velocity low amplitude) — Participants in the groups receiving DNS will be asked to hold the lower leg in the side lying position with the lower leg in the extended position and to clamp the upper leg to the lower leg with hip and knee flexion. During the application, the HLVA technique will be applied once by positioning the hypothenar part of the physiotherapist's hand on the transverse process of the lumbar vertebra where tenderness is felt by palpation and vertebral subluxation is thought to be present.
  Arms: CM + DNS Group; Chiropractic Manipulation (CM) Group
Other: Dynamic Neuromuscular Stabilization — Participants in the groups receiving DNS exercise therapy will be given individualized exercises under the supervision of a physiotherapist. First, the participants were taught posterior diaphragm activation in the supine position and the ability to direct the intraabdominal pressure caudally, while preventing the cranial movement of the thorax, so that the chest and pelvis are in a neutral position and the thoracic diaphragm and pelvis are aligned in parallel. Participants will then be taught the ability to perform a chin tuck without disturbing the alignment of the rib cage. In this way, the cervical diaphragm, thoracic diaphragm and pelvic diaphragm will be aligned in parallel. Our aim in this alignment will be to activate the deep stabilizers as a reflex response to intra-abdominal pressure change with the correct diaphragm movement pattern. Participants will be asked to focus on and maintain this alignment throughout the entire DNS exercise pattern.
  Arms: CM + DNS Group; Dynamic Neuromuscular Stabilization (DNS) Group

SUMMARY:
Our aim is to contribute to the literature by comparatively examining the effects of DNS exercises and chiropractic HVLA manipulation on pain, pain-related functional impairment (disability), physical competence level, dynamic fitness level of core muscles and postural deviations in patients with chronic nonspecific low back pain.

DETAILED DESCRIPTION:
Sixty volunteers aged between 20 and 45 years will participate in this study. Before starting the study, anthropological measurements (height, weight, body mass index) were made. After these measurements, the participants will be randomly divided into four groups.

The groups will be formed as chiropractic manipulation (CM) group (n=15), dynamic neuromuscular stabilization (DNS) group (n=15), CM + DNS group (n=15) and control group (CG) (n=15).

The KM group will receive 8 sessions of High Velocity Low Amplitude (HVLA) chiropractic manipulation twice a week for 4 weeks and the DNS group will receive 8 sessions of (DNS) exercise twice a week for 4 weeks and each session will last 50 minutes. The KM+DNS group will receive a total of 8 sessions of DNS exercises and HVLA chiropractic manipulation twice a week for 4 weeks.

Participants will be assessed a total of 3 times during the study; just before the intervention starts, 2 weeks after the intervention starts, after the 4th session, 4 weeks after completing the intervention, after the 8th session.

Participants will be assessed with Visual Analog Scale (VAS), Roland Morris Disability Questionnaire (RMDQ), Dynamic Neuromuscular Stabilization - Heel Slip Test (DNS-HS), Oswety Disability Index (ODI) and posture assessment will be performed using PostureScreen Mobile application.

ELIGIBILITY:
Inclusion Criteria:

* 7 points in Oswetry Disability Index (ODI)
* Participants should be between the ages of 20 and 45
* Normal radicular tests
* Being diagnosed with low back pain 6 months
* Not having perception problems and being able to cooperate well
* Signing the voluntary consent form

Exclusion Criteria:

* Pregnancy
* History of previous spinal canal surgery
* Presence of neurological deficits
* Presence of cancer
* Having an inflammatory or rheumatologic disease
* Spinal deformities (due to infection or trauma, compression fracture)

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | This scale will be used to subjectively assess the pain levels of the participants in the 4-week protocol; just before the beginning of the study, in the second week and in the 4th week of the study.
  The pain level of the patients will be measured with this scale. The length of the distance from the starting point of no pain to the location marked by the patient indicates the patient's pain numerically. Pain scoring according to the visual analog scale is usually graded with 0 points as no pain and 10 points as the worst pain imaginable.
Physical Adequacy Level | This scale will be used to subjectively assess the physical adequacy level of the participants in the 4-week protocol; just before the beginning of the study, in the second week and in the 4th week of the study.
  The Roland Morris Disability Questionnaire will be used to assess this parameter. This questionnaire is a subjective assessment method that evaluates the level of physical competence of individuals. The questionnaire consists of 24 items that are answered
Disability Level | This scale will be used to subjectively assess the disability levels of the participants in the 4-week protocol; just before the beginning of the study, in the second week and in the 4th week of the study.
  The Oswetry Disability Index will be used to assess the extent to which individuals' low back pain affects their daily lives and the functional status of the individual. The questionnaire, which consists of 10 questions in total, includes 6 options for each question, the options are scored between 0-5 and the sum of the scores is divided into 5 classes according to the percentile obtained by taking the percentage of the maximum score of the questionnaire.
Dynamic Stabilization and Adaptibility | This scale will be used to subjectively assess the dynamic stabilization and adaptibility levels of the participants in the 4-week protocol; just before the beginning of the study, in the second week and in the 4th week of the study.
  DNS-HS Dynamic Neuromuscular Stabilization - Heel Sliding Test will be used to measure the dynamic stabilization and adaptation level of the participants. The DNS-HS test is useful to objectively measure the dynamic adaptability of core muscles and aid in early diagnosis. It is a promising test that provides objective data that can be used to dynamically assess stabilization ability.
Posture | This mobile app will be used to assess the postural dysfunctions of the participants in the 4-week protocol; just before the beginning of the study, in the second week and in the 4th week of the study.
  PostureScreen to evaluate the posture disorders of the participants. It is a validated and reliable application designed to examine posture and present numerical data with the help of the camera system on mbil devices with Android and iOS operating systems. Participants were asked to wear appropriate clothing so that the upper body and knees remained open during the evaluation, and photographing was performed in static posture on a flat surface and in front of a flat background in front, back and both sides, leaving 3 meters between the participant and the device to be photographed fixed with a tripod. According to the reference points marked on the photograph, postural disorder values and the degree of disorder were calculated for each individual as the degree of deviation from normal posture by means of the software system in the application.

CONTACTS AND LOCATIONS:
Overall Officials: SEFA HAKTAN HATIK, Study Director — Sinop University
Locations (1):
- Sefa Haktan Haktik, Sinop, Turkey (Türkiye)